CLINICAL TRIAL: NCT00305045
Title: Treating Refractory Major Depressive Disorder With Repetitive Transcranial Magnetic Stimulation: A Double-blind, Sham-controlled, Longitudinal Study.
Brief Title: Treating Refractory Major Depressive Disorder With Repetitive Transcranial Magnetic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Z. J. Daskalakis, Director, Brain Stimulation Treatment and Research Program, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 237/2004
Record Dates: First submitted 2006-03-19; First posted 2006-03-21 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Repetitive Transcranial Magnetic Stimulation; Treatment resistance
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-frequency Left (HFL) (Active Comparator): Intensity: rTMS treatment intensity determined by using resting motor threshold (RMT). Subjects under age 65 will have treatment delivered at 100% of the RMT; those over age 65 will have treatment delivered at 120% of the RMT.
  Site of Stimulation: left hemisphere of DLPFC.
  Frequency: 10 Hz.
  Duration: 29 - 5 second trains with 30 second inter-train interval.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Bilateral (Active Comparator): Intensity: rTMS treatment intensity determined by using resting motor threshold (RMT). Subjects under age 65 will have treatment delivered at 100% of the RMT; those over age 65 will have treatment delivered at 120% of the RMT.
  Sites of Stimulation: right and left hemispheres of the DLPFC.
  Frequency: 1 Hz over the right DLPFC followed by 10 Hz over the left DLPFC.
  Duration: i) low-frequency right: 4 trains of 100 second duration and one train of 65 second duration, with a 30 second inter-train interval, followed by ii) HFL: 15 - 5 second trains with 30 second inter-train interval.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham Stimulation (Sham Comparator): Stimulation will occur over the site of active treatment, but with only the side-edge resting on the scalp. It will be administered as HFL for 17 minutes, with the coil angled 45 degrees away from the skull in a single-wing tilt position. This method produces sound and some somatic sensation (e.g., contraction of scalp muscles) similar to those of active stimulation, but with minimal direct brain effects.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Magnetic pulses to specified brain structures.
  Other Names: MagPro X100 Series (Medtronic A/S, Copenhagen, Denmark)

SUMMARY:
Studies exploring the efficacy of repetitive transcranial magnetic stimulation (rTMS) as a treatment for refractory major depressive disorder (MDD) have shown significant promise. Despite this, several questions regarding the treatment parameters needed to optimize efficacy remain. Moreover, there is also a lack of clear understanding as to the therapeutic mechanisms involved. For example, several lines of evidence suggest that patients with MDD have deficits in cortical inhibition (CI) and that these deficits are key to understanding the pathophysiology of this disorder. With this study, we seek to confirm the therapeutic potential of an acute course of rTMS for treatment-refractory MDD in a large sample of patients. In addition, we will strive to clarify the neurophysiological mechanisms through which rTMS exerts its therapeutic effects, using both TMS and electroencephalography/event related brain potential (EEG/ERP) measures of neurophysiological activity. Moreover, in this study, we intend to investigate the efficacy of a maintenance course of rTMS in an effort to prevent symptom recurrence.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is one of the most prevalent mental illnesses in North America, affecting approximately 4% of Canadians annually. Though a number of effective treatments are available, as many as 15% of those diagnosed with a depressive disorder die by suicide, 30% fail to respond to treatment and approximately 60% experience a relapse. These statistics emphasize the need to optimize treatment response, as well as to understand the neurobiological mechanisms mediating MDD, in order to improve therapeutic outcome.

To date, few alternatives have been available for the treatment of refractory symptoms - one alternative is electroconvulsive therapy (ECT); however, this treatment is associated with significant side effects, most notably memory impairment. Also, ECT requires the use of a general anesthetic, and, thus, is a relatively more invasive procedure with an increased risk of complications. In addition, the stigma associated with ECT often limits its widespread acceptance as a treatment for depressive symptoms. rTMS has been shown to be an effective therapeutic tool for the treatment of several neuropsychiatric disorders, including MDD and schizophrenia. In MDD, two types of rTMS treatment protocols have been shown to be effective. These include high frequency (10Hz) rTMS applied to the left dorsolateral prefrontal cortex (DLPFC) (HFL) and low frequency (1Hz) rTMS applied to the right DLPFC (LFR). More recently, preliminary studies combining LFR rTMS with HFL rTMS - in effect, Bilateral rTMS - have shown this method to be safe, well-tolerated, and superior to using either stimulation protocol alone. However, other studies have demonstrated equivocal efficacy of rTMS treatment for MDD. Several methodological limitations, however, have tainted most treatment studies, precluding the ability to make definitive conclusions regarding the efficacy of rTMS for MDD. These limitations include: 1) small sample sizes; 2) a lack of adequate double-blind conditions; 3) a lack of adequate treatment duration; 4) biased randomization; 5) patient heterogeneity; 6) a lack of maintenance treatment protocols; 7) an unclear understanding of the parameters necessary to optimize treatment; and 8) insufficient understanding of the neurophysiological mechanisms mediating the therapeutic efficacy of rTMS treatment.

With this study, we intend to rectify these methodological limitations by: including a large sample of treatment refractory patients, who meet pre-established criteria for treatment resistance; excluding patients with comorbid Axis II psychopathology; developing and maintaining a randomized and double-blind protocol prior to study initiation; extending active rTMS treatment courses; evaluating 2 different treatment protocols; and evaluating whether the induction of CI mediates the therapeutic effects of rTMS on depressive symptoms.

With regard to the latter objective, several lines of evidence support our hypothesis regarding a mechanistic role of CI in the therapeutic effects of rTMS. First, ECT-mediated increases in EEG slow wave activity (SWA) and cortical GABA in patients with MDD suggest that enhanced CI is related to clinical improvement. Second, MDD is a disorder that has been associated with deficits in CI. Third, deficits in CI, as indexed through cortical GABA, were rectified by supplementing antidepressant medication. In addition, a core deficit in MDD - cognitive inhibition - is conceptually related to impaired CI. Cognitive inhibition refers to the ability to ignore or inhibit mental events. Those with MDD typically experience a pronounced difficulty shifting thoughts away from negative ideas. In fact, impaired cognitive inhibition for depressogenic thoughts and information has been proposed as a mechanism and/or risk factor underlying the development and maintenance of MDD. Research in our event-related potential (ERP) lab has examined the neurophysiological correlates of CI in healthy adults and in clinical groups. During the Stroop task, CI is associated with an increased negative voltage shift peaking between 400 and 500 milliseconds over the frontocentral region of the scalp, with a decreased positivity over the left parietal region, referred to as the N450 or N500. The experimental manipulation in the present study is distinct from our ongoing MDD-ERP work in that we now have the ability to examine changes in the N450 response following anticipated rTMS-induced improvements in CI. Thus, if rTMS does bring about improvements in CI, and CI is related to cognitive inhibition, this should be associated with normalization of the N450 response in MDD.

Objectives

1. To evaluate the efficacy of an acute course of rTMS to treat patients with treatment refractory MDD.
2. To evaluate which stimulus protocol demonstrates superior therapeutic efficacy.
3. To evaluate whether the induction of CI mediates the therapeutic effects of rTMS for treatment refractory MDD.
4. To evaluate the efficacy of a maintenance course of rTMS, for those who responded to rTMS treatment, in preventing the recurrence of depressive symptoms.
5. To measure whether changes in CI are associated with changes in cognitive inhibition related to emotional information, as measured by ERP and the Emotional Stroop Task.

Hypotheses

1. In the acute treatment phase, active rTMS will be effective in treating refractory MDD compared to sham treatment.
2. Bilateral and HFL rTMS will be shown to have superior therapeutic efficacy to sham rTMS, although Bilateral rTMS will be shown to have superior therapeutic efficacy compared to HFL stimulation.
3. The induction of CI will be shown to mediate the therapeutic effects of rTMS on refractory symptoms in patients with MDD.
4. Biweekly maintenance rTMS will be effective in preventing the relapse of depressive symptoms.
5. Prior to rTMS treatment, patients will exhibit diminished neurophysiological indices of cognitive inhibition, as measured by the N450 component of the ERP. If rTMS effectively increases CI, this increase should be associated with improvements in cognitive inhibition, as measured by normalization of the N450.

ELIGIBILITY:
Inclusion Criteria:

* are voluntary and competent to consent based on their ability to provide a spontaneous narrative description of the key elements of the study (based on the MacCAT-CR)
* have a Structured Clinical Interview for DSM-IV (SCID) confirmed DSM-IV diagnosis of MDD with no co-morbid borderline personality disorder and/or antisocial personality disorder, as confirmed by the Structured Clinical Interview for DSM-IV Axis II Disorders (SCID-II)
* are between the ages of 18 and 85
* have failed to achieve a clinical response to at least 2 separate antidepressant trials of sufficient dose for at least 6 weeks, according to Stage II criteria outlined by Thase et al., or could not tolerate at least 2 trials of antidepressant medication
* have a score greater than or equal to 22 on the 17-item HAM-D
* no major, unstable medical and/or neurological conditions, such as seizures, stroke, hypertension, diabetes, coronary artery disease, thyroid problems, respiratory illness, allergies and presence of metal implants.

Exclusion Criteria:

* have a history of DSM-IV substance dependence in the last 6 months, and have DSM-IV substance abuse in the last month
* history of self-harm behaviour in past 6 months
* have a concomitant major, unstable medical or neurologic illness, or have had a history of seizures
* are acutely suicidal
* are pregnant
* have metal implants
* are currently (or in the last 4 weeks) taking: (1) more than lorazepam 2 mg daily (or equivalent); (2) monoamine oxidase inhibitors; and/or (3)bupropion due to its associated increased risk for seizures.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2005-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Degree of change on the 17-item Hamilton Rating Scale for Depression (HAM-D) | Weekly for 3 consecutive weeks. Select groups of subjects may be reassessed for an additional 3 to 52 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Zafiris J Daskalakis, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Fitzgerald PB, Brown TL, Marston NA, Daskalakis ZJ, De Castella A, Kulkarni J. Transcranial magnetic stimulation in the treatment of depression: a double-blind, placebo-controlled trial. Arch Gen Psychiatry. 2003 Oct;60(10):1002-8. doi: 10.1001/archpsyc.60.9.1002. PMID 14557145
- [Background] Klein E, Kreinin I, Chistyakov A, Koren D, Mecz L, Marmur S, Ben-Shachar D, Feinsod M. Therapeutic efficacy of right prefrontal slow repetitive transcranial magnetic stimulation in major depression: a double-blind controlled study. Arch Gen Psychiatry. 1999 Apr;56(4):315-20. doi: 10.1001/archpsyc.56.4.315. PMID 10197825
- [Background] Grunhaus L, Schreiber S, Dolberg OT, Polak D, Dannon PN. A randomized controlled comparison of electroconvulsive therapy and repetitive transcranial magnetic stimulation in severe and resistant nonpsychotic major depression. Biol Psychiatry. 2003 Feb 15;53(4):324-31. doi: 10.1016/s0006-3223(02)01499-3. PMID 12586451
- [Background] Sanacora G, Mason GF, Rothman DL, Hyder F, Ciarcia JJ, Ostroff RB, Berman RM, Krystal JH. Increased cortical GABA concentrations in depressed patients receiving ECT. Am J Psychiatry. 2003 Mar;160(3):577-9. doi: 10.1176/appi.ajp.160.3.577. PMID 12611844
- [Background] Sanacora G, Mason GF, Krystal JH. Impairment of GABAergic transmission in depression: new insights from neuroimaging studies. Crit Rev Neurobiol. 2000;14(1):23-45. doi: 10.1615/critrevneurobiol.v14.i1.20. PMID 11253954
- [Background] Sanacora G, Mason GF, Rothman DL, Krystal JH. Increased occipital cortex GABA concentrations in depressed patients after therapy with selective serotonin reuptake inhibitors. Am J Psychiatry. 2002 Apr;159(4):663-5. doi: 10.1176/appi.ajp.159.4.663. PMID 11925309
- [Derived] Trevizol AP, Goldberger KW, Mulsant BH, Rajji TK, Downar J, Daskalakis ZJ, Blumberger DM. Unilateral and bilateral repetitive transcranial magnetic stimulation for treatment-resistant late-life depression. Int J Geriatr Psychiatry. 2019 Jun;34(6):822-827. doi: 10.1002/gps.5091. Epub 2019 Apr 8. PMID 30854751
- [Derived] Weissman CR, Blumberger DM, Brown PE, Isserles M, Rajji TK, Downar J, Mulsant BH, Fitzgerald PB, Daskalakis ZJ. Bilateral Repetitive Transcranial Magnetic Stimulation Decreases Suicidal Ideation in Depression. J Clin Psychiatry. 2018 May/Jun;79(3):17m11692. doi: 10.4088/JCP.17m11692. PMID 29701939
- [Derived] Blumberger DM, Mulsant BH, Fitzgerald PB, Rajji TK, Ravindran AV, Young LT, Levinson AJ, Daskalakis ZJ. A randomized double-blind sham-controlled comparison of unilateral and bilateral repetitive transcranial magnetic stimulation for treatment-resistant major depression. World J Biol Psychiatry. 2012 Sep;13(6):423-35. doi: 10.3109/15622975.2011.579163. Epub 2011 Jul 8. PMID 21736507
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research